CLINICAL TRIAL: NCT06356402
Title: A Feasibility Study of the Investigation on the Efficacy of Oral Health Education for Mothers (OHEM) Module for Improving Oral Hygiene in Children.
Brief Title: An Investigation of the Efficacy of OHEM for Improving Oral Hygiene in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Dr.Sidra Mohiuddin, Associate Professor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8510224SMCPD
Record Dates: First submitted 2024-03-12; First posted 2024-04-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Exhibitions as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OHEM- Lecture (Experimental): In this arm, OHEM will be delivered by the lecture to the participants.
  Interventions: Behavioral: Oral Health Educational Module for Mothers (OHEM) lecture
- OHEM-Exhibition (Experimental): In this arm, OHEM will be delivered by the exhibition to the participants.
  Interventions: Behavioral: Oral Health Educational Module for Mothers (OHEM) exhibition
- OHEM-Demonstration (Experimental): In this arm, OHEM will be delivered by the demonstration to the participants.
  Interventions: Behavioral: Oral Health Educational Module for Mothers (OHEM) demonstration
- Control (No Intervention): There will be no educational intervention given to the control group. However, this group will receive oral hygiene kits and a booklet without instruction to teach their children.

INTERVENTIONS:
Behavioral: Oral Health Educational Module for Mothers (OHEM) lecture — OHEM via lecture will be delivered to the mothers by an oral health professional who will be instructed to teach their children.
  Arms: OHEM- Lecture
Behavioral: Oral Health Educational Module for Mothers (OHEM) exhibition — OHEM via exhibition will be delivered to the mothers who will be instructed to teach their children.
  Arms: OHEM-Exhibition
Behavioral: Oral Health Educational Module for Mothers (OHEM) demonstration — OHEM via demonstration will be delivered to the mothers by an oral health professional who will be instructed to teach their children.
  Arms: OHEM-Demonstration

SUMMARY:
This pilot study evaluates the feasibility of conducting a larger Randomized Controlled Trial to compare three oral health education delivery methods to a control group. Except for the control group, mothers in the three intervention groups will receive the same oral health education based on the OHEM module but differ in the delivery methods, namely lecture, exhibition, and demonstration. All groups will receive a booklet and oral hygiene kits and be instructed to educate their children at home. Pre- and post-intervention assessments include the satisfaction of participants, the researchers' evaluation and cost of the trial, oral hygiene status, and the knowledge of the parents and children.

DETAILED DESCRIPTION:
Research question:

There is lacking evidence that oral health education via family-based intervention is effective in improving oral hygiene in children.

OHEM:

A manual, the Oral Health Educational Module (OHEM), has been developed for oral health educators planning a family-based intervention to improve oral health in children by educating and empowering the mothers. OHEM aims to educate mothers about oral health and guide them to share the knowledge with their children. The content includes basic oral health knowledge and the description for preparing and delivering intervention and comes with instruments for assessing the understanding of mothers and children. Educators can choose to carry out the intervention using OHEM via three delivery methods either in a lecture, exhibition, and/or demonstration and each will present the same educational messages.

Objectives:

General objective: To investigate the feasibility of conducting a larger RCT for comparing the efficacy of the OHEM module delivered via lecture, exhibition, and demonstration to a control group.

Primary objective:

1. To determine the satisfaction of participants with the intervention program using 10 item questions relating to the organisation, researcher's attitude, recruitment process of trial, intervention process, OHEM content and delivery method, OHEM session's arrangement and venue, screening process, and fruitfulness of research among families.
2. To assess the recruitment and participation of the participants in the study.
3. To determine the cost of the trial.

Secondary objectives are:

4. To assess changes in the outcomes of the trial after the intervention in mothers and children: i) Dental plaque status ii) Gingival status iii) Oral health knowledge, attitudes, and practices iv) Oral health behaviors (tooth brushing and dental flossing skills) v) Oral health-related quality of life using OHIP-14

Methods:

Study design: This is a randomized controlled trial feasibility study comparing four groups: Lecture, Exhibition, Demonstration, and Control.

Study location: Ziauddin University Primary Health Care Center, Union Council Gulshan-e-Sikandarabad Kemari, Karachi, Pakistan. The area of Gulshan-e-Sikandarabad comprises five housing blocks.

Sample: The study participants will include mother-child dyads; the intervention is provided to the mothers and the outcomes will be assessed in the mothers and children.

Sample size: The main study assumed that children in the intervention groups would have 6.6 times greater odds of improving their gingival status one level better than before the intervention compared to the control group. Using the Open Epi sample size calculator, the sample size needed for assessing the efficacy of OHEM is n = 112 per group based on 80 % power and 5% significant level and n = 135 per group after accounting for a 20% loss to follow-up (N= 540). The present feasibility study will recruit 30% of the sample which is 41 dyad pairs per group or 164 dyad pairs in four groups.

Sampling technique: A stratified randomized sampling method to select the participants. It will randomly select, i) four of five residential blocks, and then ii) five streets from each block. Each block will be randomly assigned to one of the intervention or control groups.

The systematic random sampling technique (every second household) will be used to select a household with a mother-child dyad from each street.

Data collection:

1. Approach and explain to mothers at each identified household, assess the suitability based on the inclusion and exclusion criteria, and obtain consent.
2. Carry out baseline assessments on mothers and children. Participants will be asked to complete the questionnaires and undergo oral screening for dental plaque and gingivitis as well as assessment for behavioral skills (tooth brushing and dental flossing skills). They will be given an appointment to attend the respective intervention programs which will be carried out on separate days.
3. Mothers in the intervention groups will receive the allocated intervention, a booklet including a summary of oral health information, and an oral hygiene kit with toothbrushes, family-size toothpaste, mouthwash solution, and dental floss. They will be instructed to educate their children about oral health knowledge.

   The control group will receive only the booklet without any instruction and an oral hygiene kit. The participants will be asked not to share the details of the intervention with other participants or individuals known to be involved in the study.
4. The mothers and children will be asked to attend the post-intervention assessment after three months in which they will complete the questionnaires and undergo clinical and behavioral skill assessment.

Only one examiner (dentist) will carry out the clinical and behavioral assessments and will be blinded to the intervention group assignment.

Instrument and tools The following tools will be used to collect the data from the mother-child dyad.

i. Feasibility assessment measures:

1. Satisfaction of participants,
2. Recruitment and participation of the participants in the study,
3. Cost of the trial

ii. Dental plaque index using Silness and Loe criteria at pre- and post-intervention

iii. Gingival index using Loe and Silness criteria at pre- and post-intervention

iii. OHEM-KAP (Knowledge, attitude, practices) Questionnaire for mothers and children at pre- and post-intervention

iv. Tooth brushing and Dental flossing skills checklist at pre- and post-intervention

v. OHIP-14 (Oral health impact profile - 14) Questionnaire at pre- and post-intervention

Intervention The intervention will deliver the same knowledge content and use the same materials, but the latter can be in different forms according to the delivery method. For example, pictures of tooth anatomy will be used in all three delivery methods, a toothbrush will be shown as a picture in the lecture and the real product will be presented in the exhibition and demonstration, and toothbrushing practice will be presented as pictures/videos in the lecture and exhibition and a live demo during the demonstration.

OHEM-L: The lecture is a live talk by an educator aided by Power Point slides based on OHEM and delivered to a group of 20 participants/session for 30- to 40 minutes with no Q&A sessions.

OHEM-E: The exhibition is a display of educational posters and real exhibits based on OHEM. The participants will be given instructions to carry out self-learning by observing and reading the information. The participants will view the exhibits as they arrive but with some crowd control. The exhibition session would take 30-40 minutes to complete with no explanation by an educator and no Q&A at the end of the session.

OHEM-D: The demonstration is a live presentation by an educator with the aid of posters, actual products, and tooth models, and a live demo of toothbrushing, dental flossing, and mouth rinsing techniques based on OHEM. The demonstration will be delivered to a group of n=10 participants/ session for 30 - 40 minutes without a Q&A session.

All participants in the intervention groups will be instructed to teach their children what they have learned with the help of the booklet. Participants will also be taught how to teach their children.

Control: This group will not receive any intervention. However, they will be provided with an oral health education booklet without instructions to teach their children at home and an oral hygiene kit.

There will be no specific Q & A session for all groups. However, to keep the trial pragmatic and encourage a knowledge-seeking attitude among the mothers, the educator will respond to the queries if participants have any and including facilitating with hands-on practice.

ELIGIBILITY:
The inclusion criteria of the study are based on mothers and children.

Inclusion criteria for Mothers:

1. Mothers with children aged 12 to 15 years old, who are residing in Gulshan-e-Sikandarabad with no plan to move within the next 12 months.
2. Mothers with the ability to understand and read the Urdu language.
3. Only biological mothers with good physical and psychological health.

Exclusion criteria for mothers:

1. Mothers with new-born
2. Mothers with a history of receiving formal oral health promotion or preventive programs.

Inclusion criteria for Children:

1. Aged 12,13,14, and 15 years old (studying in classes 6,7,8, and 9 respectively) residing in union council Gulshan-e-Sikandrabad,
2. Live with biological mothers at home,
3. Present with moderate to severe plaque accumulation and gingivitis during oral screening.

Exclusion criteria for Children:

1. Have genetic or medical conditions, such as physical and psychological disabilities that can affect the comprehension of instruction and tooth brushing activities, such as learning disabilities or auditory or visual disorders.
2. Have genetic dental anomalies such as anodontia, amelogenesis imperfecta, and supernumerary teeth.
3. Have been previously exposed to any form of oral health education.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of participants: | six months
  i. Are you satisfied with the program's organisation? ii. Are you satisfied with the researcher's attitude during the trial? iii. Are you satisfied with the recruitment process? iv. Are you satisfied with the intervention process? v. Are you satisfied with the content taught during the intervention? vi. Are you satisfied with the researcher's delivery of the content? vii. Are you satisfied with arranging the OHEM sessions at the venue? viii. Is the environment at the venue conducive to learning? ix. Are you satisfied with the baseline and final stage of the oral screening process? x. Do you trust the researcher that her research will be fruitful for you and your family? The satisfaction will be assessed using a 10-item questionnaire mentioned in the primary objective. Participants will respond to each question using a 5-point Likert scale rating; each item will be reported as the percentage of participants who are at least somewhat satisfied (score 3,4,5)
Recruitment and participation of participants in the study | six months
  i) How well participants cooperated
  1. During the recruitment/baseline data collection
  2. During the intervention
  3. During the follow-up/ final data collection process
  Additional comments by the researcher:______________________
  The recruitment will be assessed on a Likert scale rating (very dissatisfied, dissatisfied, somewhat satisfied, satisfied, very satisfied); each item will be reported as the percentage of participants who are at least somewhat satisfied (score 3,4,5), whereas the participation of the participants will be assessed in percentage.
Cost of the trial | six months
  The cost of the trial will be assessed by comparing the cost of the expenditure at the end of the trial. i) Travelling cost, ii) Preparation of materials for the OHEM lecture, exhibition, and demonstration session cost, iii) Conducting the OHEM lecture, exhibition, and demonstration sessions cost, iv) Cost of the incentives for the participants, v) Cost for the volunteers of the trial.

SECONDARY OUTCOMES:
Dental plaque scores | six months
  Change in dental plaque scores among mothers and children between intervention and control groups, assessed pre- and post-intervention, using mean and Standard Deviation; lower scores will indicate good oral hygiene.
Gingival scores | six months
  Change in gingival scores among mothers and children between intervention and control groups, assessed pre- and post-intervention, using mean and Standard Deviation; lower scores will indicate good oral hygiene.
Oral health KAP scores | six months
  Change in oral health KAP scores among mothers and children between intervention and control groups, assessed pre and post-intervention, using mean and Standard Deviation; the higher scores indicate better KAP.
Oral health behaviors | six months
  Change in skills (tooth brushing and dental flossing) among mothers and children between intervention and control groups, assessed pre- and post-intervention, using add scores; higher scores indicate good behaviours.
Oral health-related quality of life using Oral health impact profile-14 | six months
  Change in oral health impact profile-14 among mothers and children between intervention and control groups, assessed pre- and post-intervention, using add scores and mean and Standard Deviation; higher scores indicating poor oral health.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Mohiuddin, MDS, Principal Investigator — Ziauddin University
Locations (1):
- Primary Healthcare Center Gulshan-e-Sikandarabad Shireen Jinnah Colony, Karachi, Pakistan

REFERENCES:
- [Background] Yusoff M. S. B. ABC of content validation and content validity index calculation. J Education in Medicine Journal. 2019;11(2), 49-54.
- [Background] World Health Organization. Oral health surveys: basic methods: World Health Organization. 2013.
- [Background] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Silveira M. F., Pinho L. d. & Brito M. F. S. F. Validity and reliability of the oral health impact profile instrument (OHIP-14) in adolescents. J Paidéia. 2019;29.
- [Background] Crews K, O'Hara J, Gordy F, Penton N. The Bass technique: Charles Cassidy Bass' legacy. Miss Dent Assoc J. 1995 Summer;51(2):18-20. PMID 9569849
- [Background] Newman M. G., Takei H., Klokkevold P. R. & Carranza F. A. Carranza's Clinical Periodontology: Elsevier health sciences. 2011.
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Saied-Moallemi Z, Virtanen JI, Ghofranipour F, Murtomaa H. Influence of mothers' oral health knowledge and attitudes on their children's dental health. Eur Arch Paediatr Dent. 2008 Jun;9(2):79-83. doi: 10.1007/BF03262614. PMID 18534175